CLINICAL TRIAL: NCT01578148
Title: Noxipoint Therapy vs. Standard Physical Therapy Using Electrical Stimulation for Chronic Pain
Brief Title: Noxipoint Therapy Versus Standard Physical Therapy Using Electrical Stimulation for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pain Cure Center, California (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NT-01-2012
Record Dates: First submitted 2012-04-13; First posted 2012-04-16 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Shoulder Pain; Neck Pain
Keywords: Cervical pain; Cervicalgia,; Cervicodynia; Neck ache; Neckache; Shoulder pain; Shoulder impingement syndrome
MeSH Terms: conditions — Shoulder Pain; Neck Pain; Shoulder Impingement Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Noxipoint Therapy (Experimental)
  Interventions: Procedure: Noxipoint Therapy
- Physical Therapy (Active Comparator)
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Procedure: Noxipoint Therapy — Patients will be treated with a TENS device, following Noxipoint Therapy guidelines:
  1. Find the cause of the pain via Noxipoint: For each injured muscle/tissue, it is discovered that there are always a pair of points at the skin surface locations of its nociceptors that are painful at light press (named "Noxipoints").
  2. Stimulate the corresponding pair of Nocipoints following a narrowly defined combination of intensity/ frequency (inducing the C-fiber response) and duration (about 1.5-3 minutes) of TENS at the two targeted Noxipoints.
  3. Repeat (a) to (b) above for each identified injured muscle group until all pain areas are eliminated or when the session time is up.
  4. Instruct the subject not to use the newly recovered muscle/tissue too much an estimated rest period depending on his/her age.
  Other Names: Koo's Pain Cure Therapy
  Arms: Noxipoint Therapy
Procedure: Physical Therapy — The 1.5-hour physical therapy in the control arm are provided both as standard of care and sham device comparison to Nocipoint Therapy, following these guidelines:
  1. TENS stimulation (45 minutes):
     • Electrodes will be placed around the patient-identified general pain area on the neck /shoulder for TENS. Rotate the electrode pads around the pain area and stimulate again.
  2. Other modalities of PT per the therapist's choice:
     * Infrared treatment on the pain areas (about 15 minutes)
     * Manual therapy to cervical and/or rotator cuff areas (about 15 minutes).
     * Exercise and training:
       * Neck exercises: Range of motion exercises to include foraminal opening for about 15 minutes, and/or
       * Shoulder exercise: Range of motion exercises to include walking the arm on the wall, rotation of the upper arm for about 15 minutes
     * Hot/cold pack to the pain area for about 15 minutes
  Other Names: PT
  Arms: Physical Therapy

SUMMARY:
The purpose of this study is to validate the efficacy of Noxipoint(TM) therapy on chronic pain, and compare it with standard physical therapy using electrical stimulation on patients with chronic pain.

Invented by Dr. Charlie Koo at Stanford University, Noxipoint Therapy is a specific procedure with precise location, duration and intensity of TENS stimulation within the general FDA guidelines. The therapy substantially relieves general muscular/tendon pain and persistently restores the muscle and tendon function. The surface locations of nociceptors at the free nerve ending (i.e., "Noxipoints") are focused on in the stimulation therapy. Multiple clinical uses of Noxipoint Therapy confirmed the consistent efficacy of such stimulation at Noxipoints. An observational study of Noxipoint therapy within the FDA-approved use of TENS demonstrated an encouraging 93% success rate in eliminating the chronic pain, such as frozen shoulder pain, within 2-3 sessions. It is an order-of-magnitude improvement over the non-specific application of TENS and any other modalities in pain treatment. A unique neuro-immuno-signaling pathway that implicates the activation of adult stem cells, such as satellite cells in muscles, is implicated based on such a high success rate.

DETAILED DESCRIPTION:
View http://paincurecenter.com/Clinical_Outcome.html for the observational study mentioned in the Brief Summary above. For more detailed cases, please view http://paincurecenter.com/uploads/Nocipoint_therapy_clinical_study_w_o_ID_2011-2012.pdf

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old male or female
* Having chronic pain (ICD-9: 338.21, 338.29) in the neck/upper back (ICD-9: 723.1), or the shoulder (ICD-9: 719.41)
* Pain duration over 6 months, with at least one month of history of other therapy treatments (Physical therapy, steroid injection, acupuncture, analgesic medicine, and/or massage therapy)

Exclusion Criteria:

* Patients with BPI Severity at its Worst below 5
* Traumatic injury from external impact force
* Pain caused by traumatic bone fractures
* History of traumatic cervical injury
* History of osteoporosis
* Pain related to systemic inflammatory conditions including polymyalgia rheumatic, systemic lupus erythematosis
* Signs of psychosomatic illness
* Severe rheumatoid arthritis undergoing active treatment including DMARD biologics
* Steroid injection on pain site within 4 weeks
* Language and/or cognitive inability to complete the assessment questionnaires
* Previous TENS for pain relief
* For safety reasons, patients wearing cardiac pace makers, implanted defibrillator, or pregnant women

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) Severity of the Pain at Its Worst | One year
  BPI will be evaluated as the score change from the baseline. As a supplemental measure, the baseline of individual patients will also be normalized to 100%, with the change being a percentile of the baseline.

SECONDARY OUTCOMES:
BPI Severity of the pain in the other three occasions | One year
  Besides the Severity of the Pain at Its Worst, there are three other pain measures in BPI. This measure will be used as a supporting measure fo the Primary Measure.
BPI Interference of Function | One year
  This measure is used to indicate the impact of the subject's quality of life. However, the standard questions include the therapy's functional impact on walking, which is not likely to be influenced by neck/shoulder pains in any case and thus may not be relevant. Thus, a supplemental measure excluding the impact on walking will be provided as a supplemental observation.
Range of motion | One year
  This measure will be taken whenever possible.
Shoulder Pain and Disability Index (SPADI) | One year
  SPADI will be taken from shoulder pain patients whenever possible. This is optional.
Neck Disability Index (NDI) | One year
  NDI will be taken from neck pain patients whenever possible. This is optional.

CONTACTS AND LOCATIONS:
Overall Officials: Charles C Koo, PhD, Study Director — Pain Cure Center; Charles C Koo, PhD, Principal Investigator — Pain Cure Center; David Lewis, MD, Principal Investigator — Stanford University
Locations (1):
- Pain Cure Center, Palo Alto, California, United States